CLINICAL TRIAL: NCT04482036
Title: The MObile AssessMENT of Behavioral and Psychological Symptoms of Dementia in Amnestic Mild Cognitive Impairment and Alzheimer's Disease (MOMENT) Study: A Randomized Controlled Trial
Brief Title: The MObile AssessMENT of Behavioral and Psychological Symptoms of Dementia in Amnestic MCI and AD (MOMENT) Study
Acronym: MOMENT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Principle Investigator changed careers and relinquished their NIA funded career development award, which funded the MOMENT Study. Career development awards are not transferable. Thus, the study was terminated prematurely.
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Chris Callahan, MD, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1907055854; 1K23AG059914-01A1 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-07-22 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease; Mild Memory Disturbance; Mild Cognitive Impairment
Keywords: Patient Distress; Caregiver Burden; Caregiver Stress; Mobile Phone Application; Psychological Symptoms; Behavioral Symptoms; Behavioral and Psychological Symptoms of Dementia; Neuropsychiatric Symptoms; mHealth; Mobile Health
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Caregiver Burden; Behavioral Symptoms; Behavior

STUDY DESIGN:
Intervention Model Description: The study design includes six 1-month periods. Those in the intervention group will be nested in a 2 x 6 cross-over design in which they will be randomly assigned to start with 1 of 2 schedules of Ecological Momentary Assessment (EMA) surveillance frequency (1) weekly or (2) monthly. The intervention participants will then cross-over at the end of each and every month to the other surveillance frequency condition, over a 6-month time horizon.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator will be masked to arm allocation of participants. The outcomes assessor at time of 3 month and 6 month (final) assessment will also be masked to the allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dementia Collaborative Care (Placebo Comparator): Patient and caregivers assigned to the three in-person assessments and no mobile application group will complete the following:
  * The caregiver will be asked to complete three in-person assessments that involve answering survey questions and an interview.
  * Some of the questions asked will be related to Behavioral and/or Psychological Symptoms the patient experiences.
  * The caregiver will be asked to answer questions about the patient, the patient's experience with the research study and the caregiver's own experience with the research study.
  * If the patient's "symptoms" or the caregiver's "distress" answers reach a high enough level, a member of the research study team and clinical team will contact the caregiver to ask more questions and check in on the patient and caregiver's safety.
  * The research study team will also notify Dr. Bateman (the person responsible for the research).
  Interventions: Other: Standard Assessments
- Dementia Collaborative Care Plus BrainCare Notes Application (Active Comparator): Patient and caregivers assigned to the three in-person assessments and mobile application group will complete the same tasks that Group 1 (control group) will complete with the addition of the following:
  * The caregiver will be asked to monitor the patient and complete 5 to 10-minute long surveys (the neuropsychiatric inventory questionnaire) sent to the caregiver through the mobile application or in-person at each follow-up visit.
  * The caregiver will be asked to monitor and complete these surveys at different times for a period of 6 months.
  Interventions: Other: Mobile Phone Application Assessments; Other: Standard Assessments

INTERVENTIONS:
Other: Mobile Phone Application Assessments — The BrainCare Notes app was designed to be installed on the caregiver's phone. It has the capacity to send Neuropsychiatric Inventory Questionnaire (NPI-Q) assessments to the caregiver. If the answers to the behavioral and psychological symptoms rise above the threshold, the clinicians will be notified, and a care plan will be enacted, in order to keep the patient and caregiver safe.
  The application also has the ability to send and receive private messages between caregiver and the patient's clinical care team.
  Other Names: BrainCare Notes app
  Arms: Dementia Collaborative Care Plus BrainCare Notes Application
Other: Standard Assessments — The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.

SUMMARY:
The purpose of this research study is to learn whether it is possible and useful for caregivers to report behavioral or psychological symptoms of people with mild memory problems or Alzheimer's disease through a smartphone mobile application. The investigators believe that monitoring these symptoms and having a tool, like a mobile application, can provide quicker accessibility to the patient's clinical care team, which could improve care for patients and caregivers.

These types of symptoms found in patients with mild memory problems or Alzheimer's disease are any type of psychiatric symptoms or abnormal behaviors one might develop as the result of these brain illnesses. Examples of psychological and behavioral symptoms are depression, anxiety, insomnia, irritability, agitation, and hallucinations. These symptoms differ from regular psychiatric symptoms, because they are caused by mild memory problems or Alzheimer's disease (AD). These symptoms can cause a lot of distress for patients and caregivers, and can lead to greater use of healthcare services.

DETAILED DESCRIPTION:
As a part of this research study the patient and caregiver will undergo randomization, "like flipping a coin", to assign the patient and caregiver to one of two research study groups. The patient and the partnered caregiver will join the same group. The group will either receive: 1) three in-person assessments on symptoms and behaviors that the patient may experience and a mobile application that will send surveys to the caregiver in order to rate the presence, severity and stress caused by these symptoms and behaviors; or 2) three in-person assessments on symptoms and behaviors that the patient may experience and no mobile application. The outcomes of these surveys and assessments will then be shared with the patient's clinical team.

If the caregiver is assigned to the group that receives the mobile application they will receive the surveys either weekly or monthly. After each month of completing the surveys, the frequency will change. Depending on feedback from the first 10 participants, the investigators may modify the survey rate to happen more than weekly.

ELIGIBILITY:
Inclusion Criteria:

* The patient:

  * Has Alzheimer's Disease (AD) or Amnestic Mild Cognitive Impairment (aMCI), is a Healthy Aging Brain Center, Eskenazi Health patient
  * Community dwelling
  * Has a legally authorized representative when they lack capacity to consent
* The caregiver:

  * 18 or older
  * No visual impairment
  * Community dwelling
  * Reports seeing patient most days of the week

Exclusion Criteria:

* The patient:

  * History of mental illness (Schizoaffective disorder, schizophrenia, bipolar)
  * Participating in another study
  * The potential participant with a diagnosis of either aMCI or AD communicates observable dissent.
* The caregiver:

  * History of mental illness (Schizoaffective disorder, schizophrenia, bipolar)
  * Participating in another study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Bateman, MD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dementia Collaborative Care - Patients; Dementia Collaborative Care - Caregivers: Patient and caregivers assigned to the three in-person assessments and no mobile application group will complete the following:
  * The caregiver will be asked to complete three in-person assessments that involve answering survey questions and an interview.
  * Some of the questions asked will be related to Behavioral and/or Psychological Symptoms the patient experiences.
  * The caregiver will be asked to answer questions about the patient, the patient's experience with the research study and the caregiver's own experience with the research study.
  * If the patient's "symptoms" or the caregiver's "distress" answers reach a high enough level, a member of the research study team and clinical team will contact the caregiver to ask more questions and check in on the patient and caregiver's safety.
  * The research study team will also notify Dr. Bateman (the person responsible for the research).
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
- Dementia Collaborative Care Plus BrainCare Notes Application - Patients; Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers: Patient and caregivers assigned to the three in-person assessments and mobile application group will complete the same tasks that Group 1 (control group) will complete with the addition of the following:
  * The caregiver will be asked to monitor the patient and complete 5 to 10-minute long surveys (the neuropsychiatric inventory questionnaire) sent to the caregiver through the mobile application or in-person at each follow-up visit.
  * The caregiver will be asked to monitor and complete these surveys at different times for a period of 6 months.
  Mobile Phone Application Assessments: The BrainCare Notes app was designed to be installed on the caregiver's phone. It has the capacity to send Neuropsychiatric Inventory Questionnaire (NPI-Q) assessments to the caregiver. If the answers to the behavioral and psychological symptoms rise above the threshold, the clinicians will be notified, and a care plan will be enacted, in order to keep the patient and caregiver safe.
  The application also has the ability to send and receive private messages between caregiver and the patient's clinical care team.
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
Period: Overall Study
Arm/Group | Dementia Collaborative Care - Patients | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Patients | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Started | 5 | 5 | 5 | 5
Completed | 2 | 2 | 0 | 0
Not Completed | 3 | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dementia Collaborative Care - Patients | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Patients | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 0 | 2 | 5
  >=65 years | 5 | 2 | 5 | 3 | 15
Age, Continuous [Mean (Full Range); unit: years] | 78.2 [68 to 87] | 64.4 [45 to 88] | 78.2 [70 to 84] | 70.6 [43 to 85] | 72.85 [43 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 3 | 13
  Male | 1 | 1 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 5 | 5 | 4 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Caregivers Who Completed Neuropsychiatric Interview Questionnaire (NPI-Q) at 3 Months
Time Frame: Calculated at 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Control - Dementia Collaborative Care - Caregivers: Patient and caregivers assigned to the three in-person assessments and no mobile application group will complete the following:
  * The caregiver will be asked to complete three in-person assessments that involve answering survey questions and an interview.
  * Some of the questions asked will be related to Behavioral and/or Psychological Symptoms the patient experiences.
  * The caregiver will be asked to answer questions about the patient, the patient's experience with the research study and the caregiver's own experience with the research study.
  * If the patient's "symptoms" or the caregiver's "distress" answers reach a high enough level, a member of the research study team and clinical team will contact the caregiver to ask more questions and check in on the patient and caregiver's safety.
  * The research study team will also notify Dr. Bateman (the person responsible for the research).
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
- Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers: Patient and caregivers assigned to the three in-person assessments and mobile application group will complete the same tasks that Group 1 (control group) will complete with the addition of the following:
  * The caregiver will be asked to monitor the patient and complete 5 to 10-minute long surveys (the neuropsychiatric inventory questionnaire) sent to the caregiver through the mobile application or in-person at each follow-up visit.
  * The caregiver will be asked to monitor and complete these surveys at different times for a period of 6 months.
  Mobile Phone Application Assessments: The BrainCare Notes app was designed to be installed on the caregiver's phone. It has the capacity to send Neuropsychiatric Inventory Questionnaire (NPI-Q) assessments to the caregiver. If the answers to the behavioral and psychological symptoms rise above the threshold, the clinicians will be notified, and a care plan will be enacted, in order to keep the patient and caregiver safe.
  The application also has the ability to send and receive private messages between caregiver and the patient's clinical care team.
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
Arm/Group | Control - Dementia Collaborative Care - Caregivers | Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 3 | 4
Participants | 3 | 4

2. Primary Outcome: Number of Caregivers Who Completed the Neuropsychiatric Interview Questionnaire (NPI-Q) at 6 Months
Time Frame: Calculated at 6 months
Population: The study was terminated before other participants reached the 6 month time point. Two caregivers reached the 6 month time point.
Measure: Number; unit: participants
Arm/Group | Control - Dementia Collaborative Care - Caregivers | Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
participants |  | 2

3. Primary Outcome: Number of Caregivers Who Completed the BrainCare Notes (BCN) App - Survey Burden Mean at 3 Months
Description: Randomized participants are prompted to answer the survey burden question after completion of each BCN app prompted survey. The caregivers in the control group, "Dementia Collaborative Care- Caregivers" did not utilize the BrainCare Notes application.
Time Frame: Calculated at 3 months
Population: This outcome measure is designated only to participants in the randomized group, therefore there are zero participants in the control group that completed this survey. There were only 4 randomized participants who reached this time point before the study was terminated.
Measure: Count of Participants; unit: Participants
Groups:
- Control- Dementia Collaborative Care - Caregivers: Patient and caregivers assigned to the three in-person assessments and no mobile application group will complete the following:
  * The caregiver will be asked to complete three in-person assessments that involve answering survey questions and an interview.
  * Some of the questions asked will be related to Behavioral and/or Psychological Symptoms the patient experiences.
  * The caregiver will be asked to answer questions about the patient, the patient's experience with the research study and the caregiver's own experience with the research study.
  * If the patient's "symptoms" or the caregiver's "distress" answers reach a high enough level, a member of the research study team and clinical team will contact the caregiver to ask more questions and check in on the patient and caregiver's safety.
  * The research study team will also notify Dr. Bateman (the person responsible for the research).
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
Arm/Group | Control- Dementia Collaborative Care - Caregivers | Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 4
Participants | 0 | 4

4. Primary Outcome: Number of Participants Who Completed the BrainCare Notes (BCN) App - Survey Burden Mean at 6 Months
Description: as for outcome 3
Time Frame: Calculated at 6 months
Population: This outcome measure is designated only to participants in the randomized group, therefore there are zero participants in the control group that completed this survey. There were only two randomized participants that reached the 6 month time point before the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Dementia Collaborative Care - Caregivers | Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

5. Primary Outcome: Number of Participants Who Completed the System Usability Scale (SUS) at the 3 Month Timepoint
Description: The System Usability Scale will be used to assess usability of the BrainCare Notes app at 3 months. Only the randomized participants will be completing this survey. The scale is as follows: Strongly Disagree-1, Disagree- 2, Neutral- 3, Agree- 4, Strongly Agree- 5
Time Frame: Measured at 3 months
Population: This outcome measure is designated only to participants in the randomized group, therefore there are zero participants in the control group that completed this survey. The study was terminated before the other participant reached the 3 month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Dementia Collaborative Care - Caregivers | Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 4
Participants |  | 4

6. Primary Outcome: Number of Participants Who Completed the System Usability Scale (SUS) at the 6 Month Timepoint.
Description: The System Usability Scale (SUS) will be used to assess usability of the BrainCare Notes app at 6 months. Only the randomized participants will be completing this survey. The scale is as follows: Strongly Disagree-1, Disagree- 2, Neutral- 3, Agree- 4, Strongly Agree- 5
Time Frame: Measured at 6 months
Population: This outcome measure is designated only to participants in the randomized group, therefore there are zero participants in the control group that completed this survey. The study was terminated before other participants reached the 6 month time point. Two caregivers reached the 6 month time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Dementia Collaborative Care - Caregivers | Randomized - Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
Participants |  | 2

7. Secondary Outcome: Outcome of the Change in Behavioral and Psychological Symptoms (BPSD) Score- Specifically Any Change Seen at 3 Months From What Was Reported at Baseline.
Description: The NPI-Q is a questionnaire administered to a caregiver who cares for a person with mild cognitive impairment (MCI), Alzheimer's disease (AD) or dementia.
  Symptom severity scores for each of the symptom domain range between 0-not present, 1 - mild, 2-moderate, 3-severe. The summation of all symptom severity scores have a range of a minimum score of 0 and maximum score of 36, where the higher the number indicates worse symptom severity.
Time Frame: Calculated at 3 months
Population: There were 2 patients from the control group (dementia collaborative care arm) that passed away before the 3 month period was met, therefore the outcome wasn't collected from the caregivers.
  The study was terminated before the other participant reached the 3 month time point.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 3 | 4
score on a scale | 0.33 [-4 to 7] | 1 [-7 to 8]

8. Secondary Outcome: Outcome of the Change in Behavioral and Psychological Symptoms (BPSD) Score- Specifically Any Change Seen at 6 Months From What Was Reported at Baseline.
Description: as for outcome 7
Time Frame: Calculated at 6 months
Population: The study was terminated before the other participants were able to complete this survey at the 6 month time point.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
score on a scale |  | 6 [2 to 10]

9. Secondary Outcome: Outcome of the Change in Caregiver Distress Score- Specifically Any Change Seen at 3 Months From What Was Reported at Baseline.
Description: The NPI-Q is a questionnaire administered to the caregiver who cares for a person with mild cognitive impairment (MCI), Alzheimer's disease (AD) or dementia.
  The Caregiver Distress scores for each of the symptom domain range between: 0 = Not distressing at all, 1 = Minimal, 2 = Mild, 3 = Moderate, 4 = Severe, 5 = Extreme or Very Severe. The summation of all the Caregiver Distress scores ranges from a min score of 0 and max score of 60, where the higher the number indicates worse Caregiver Distress severity.
Time Frame: Calculated at 3 months
Population: There were 2 patients from the control group (dementia collaborative care arm) that passed away before the 3 month period was met, therefore the outcome wasn't collected from the caregivers. Data from the remaining participants wasn't collected as the study was terminated before reaching this time point.
  The study was terminated before the other participant reached the 3 month time point.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 3 | 4
score on a scale | 0.33 [-4 to 7] | 4.25 [-11 to 14]

10. Secondary Outcome: Outcome of the Change in Caregiver Distress Score- Specifically Any Change Seen at 6 Months From What Was Reported at Baseline.
Description: as for outcome 9
Time Frame: Calculated at 6 months
Population: The study was terminated before other participants reached the 6 month time point. Only two caregivers reached the 6 month time point.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
score on a scale |  | -3.5 [-9 to 2]

11. Other Pre Specified Outcome: Outcome of the Change in the Perceived Stress Scale 14 (PSS-14) Score- Specifically Any Change Seen at 3 Months From What Was Reported at Baseline.
Description: The PSS-14 is a validated self-reported questionnaire comprised of 14 items designed to assess stress and coping. Participants rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4" Very often." Total scores range from 0 to 56 with a higher score indicating greater perceived stress.
Time Frame: Calculated at 3 months
Population: There were 2 patients from the control group (dementia collaborative care arm) that passed away before the 3 month period was met, therefore the outcome wasn't collected from the caregivers. Data from the remaining participants wasn't collected because the study was terminated.
  The study was terminated before the other participant reached the 3 month time point.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 3 | 4
score on a scale | -1 [-7 to 6] | -3.67 [-6 to -1]

12. Other Pre Specified Outcome: Outcome of the Change in the Perceived Stress Scale 14 (PSS-14) Score- Specifically Any Change Seen at 6 Months From What Was Reported at Baseline.
Description: as for outcome 11
Time Frame: Calculated at 6 months
Population: The study was terminated before other participants reached the 6 month time point. Only two caregivers reached the 6 month time point, data from the remaining participants wasn't collected.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
score on a scale |  | 3 [1 to 5]

13. Other Pre Specified Outcome: Outcome of the Change in the Zarit Burden Interview (ZBI-12) Score- Specifically Any Change Seen at 3 Months From What Was Reported at Baseline.
Description: The ZBI-12 is a validated, caregiver self-report measure comprised of 12 items designed to assess caregiver burden in those who care for patients with advanced illness, including dementia. Participants rate items on a 5-point Likert scale, ranging from, "0 - Never" to "4 - Nearly Always." Total scores range from 0 to 48 with a higher score indicating greater caregiver burden.
Time Frame: Calculated at 3 months
Population: There were 2 patients from the control group (dementia collaborative care arm) that passed away before the 3 month period was met, therefore the outcome wasn't collected from the caregivers. Data from the remaining participants wasn't collected as the study was terminated before the time point was reached.
  The study was terminated before the other participant reached the 3 month time point.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Dementia Collaborative Care: Patient and caregivers assigned to the three in-person assessments and no mobile application group will complete the following:
  * The caregiver will be asked to complete three in-person assessments that involve answering survey questions and an interview.
  * Some of the questions asked will be related to Behavioral and/or Psychological Symptoms the patient experiences.
  * The caregiver will be asked to answer questions about the patient, the patient's experience with the research study and the caregiver's own experience with the research study.
  * If the patient's "symptoms" or the caregiver's "distress" answers reach a high enough level, a member of the research study team and clinical team will contact the caregiver to ask more questions and check in on the patient and caregiver's safety.
  * The research study team will also notify Dr. Bateman (the person responsible for the research).
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
- Dementia Collaborative Care Plus BrainCare Notes Application: Patient and caregivers assigned to the three in-person assessments and mobile application group will complete the same tasks that Group 1 (control group) will complete with the addition of the following:
  * The caregiver will be asked to monitor the patient and complete 5 to 10-minute long surveys (the neuropsychiatric inventory questionnaire) sent to the caregiver through the mobile application or in-person at each follow-up visit.
  * The caregiver will be asked to monitor and complete these surveys at different times for a period of 6 months.
  Mobile Phone Application Assessments: The BrainCare Notes app was designed to be installed on the caregiver's phone. It has the capacity to send Neuropsychiatric Inventory Questionnaire (NPI-Q) assessments to the caregiver. If the answers to the behavioral and psychological symptoms rise above the threshold, the clinicians will be notified, and a care plan will be enacted, in order to keep the patient and caregiver safe.
  The application also has the ability to send and receive private messages between caregiver and the patient's clinical care team.
  Standard Assessments: The caregiver and patient will receive the same questionnaires and surveys that the intervention group will receive. However, they will not receive the mobile phone application questionnaires.
Arm/Group | Dementia Collaborative Care | Dementia Collaborative Care Plus BrainCare Notes Application
Number analyzed (Participants) | 3 | 4
score on a scale | 1 [-5 to 8] | 0 [-6 to 5]

14. Other Pre Specified Outcome: Outcome of the Change in the Zarit Burden Interview (ZBI-12) Score- Specifically Any Change Seen at 6 Months From What Was Reported at Baseline.
Description: as for outcome 13
Time Frame: Calculated at 6 months
Population: as for outcome 12
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
Number analyzed (Participants) | 0 | 2
score on a scale |  | -1 [-2 to 0]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dementia Collaborative Care - Patients | Dementia Collaborative Care - Caregivers | Dementia Collaborative Care Plus BrainCare Notes Application - Patients | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dementia Collaborative Care - Patients (N=5) | Dementia Collaborative Care - Caregivers (N=5) | Dementia Collaborative Care Plus BrainCare Notes Application - Patients (N=5) | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers (N=5)
Hospitalization (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Bilateral pulmonary embolism
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dementia Collaborative Care - Patients (N=5) | Dementia Collaborative Care - Caregivers (N=5) | Dementia Collaborative Care Plus BrainCare Notes Application - Patients (N=5) | Dementia Collaborative Care Plus BrainCare Notes Application - Caregivers (N=5)
Pacemaker insertion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated [The Principle Investigator changed careers and relinquished their NIA funded career development award, which funded the MOMENT Study. Career development awards are not transferable. Thus, the study was terminated prematurely.]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT04482036/Prot_SAP_000.pdf